CLINICAL TRIAL: NCT03819179
Title: The Influence of Personal Care Products on the Skin Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1161875
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Microbiome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Serum (Experimental): Burt's Bees Serum
  Interventions: Other: Burt's Bees Serum
- Serum with Biulin (Experimental): Burt's Bees Serum with Biulin
  Interventions: Other: Burt's Bees Serum with Biulin
- Serum with Berenew Complex (Experimental): Burt's Bees Serum with Berenew Complex
  Interventions: Other: Burt's Bees Serum with Berenew Complex
- Serum with Ecoskin (Experimental): Burt's Bees Serum with Ecoskin
  Interventions: Other: Burt's Bees Serum with Ecoskin
- Serum with Bonicell (Experimental): Burt's Bees Serum with Bonicell
  Interventions: Other: Burt's Bees Serum with Bonicell

INTERVENTIONS:
Other: Burt's Bees Serum — This is a commercially available over-the-counter product. Ingredients: Caprylic/ Capric Trigylceride, Isopropyl Palmitate, Sweet Almond Oil, Lanette O, Water, Cetearyl Glucoside, Gluconolactone ans Sodium Benzoate, Water, Glycerin, Xanthan GUM, Tocopherol.
  Arms: Serum
Other: Burt's Bees Serum with Biulin — This is a commercially available over-the-counter product. Ingredients: Caprylic/ Capric Trigylceride, Isopropyl Palmitate, Sweet Almond Oil, Lanette O, Water, Cetearyl Glucoside, Gluconolactone ans Sodium Benzoate, Water, Glycerin, Xanthan GUM, Tocopherol, PreBIULIN FOS (GOVA).
  Arms: Serum with Biulin
Other: Burt's Bees Serum with Bonicell — This is a commercially available over-the-counter product. Ingredients: Caprylic/ Capric Trigylceride, Isopropyl Palmitate, Sweet Almond Oil, Lanette O, Water, Cetearyl Glucoside, Gluconolactone ans Sodium Benzoate, Water, Glycerin, Xanthan GUM, Tocopherol, Bonicel (Ganaden).
  Arms: Serum with Bonicell
Other: Burt's Bees Serum with Berenew Complex — This is a commercially available over-the-counter product. Ingredients: Caprylic/ Capric Trigylceride, Isopropyl Palmitate, Sweet Almond Oil, Lanette O, Water, Cetearyl Glucoside, Gluconolactone ans Sodium Benzoate, Water, Glycerin, Xanthan GUM, Tocopherol, BeRenew CLR Complex (CLR).
  Arms: Serum with Berenew Complex
Other: Burt's Bees Serum with Ecoskin — This is a commercially available over-the-counter product. Ingredients: Caprylic/Capric Triglyceride, Dimer Dilinoleyl Dimer Dilionoleatem, Silica, Citronellyl Methylcrotonate, Tocopheryl Acetate, Xymenynic Acid, Alpha-glucan Oligosaccharide, Fragrance, Slareolide, Polymnia sonshifolia root juice, Helianthus annuus (sunflower) seed oil, Maltodextrin, Tocopherol, Beta-sitosterol, Lactobacillus, Squalene.
  Arms: Serum with Ecoskin

SUMMARY:
To evaluate whether personal care products shift the skin microbiome bacteria and diversity after a week of daily use.

DETAILED DESCRIPTION:
Studies have shown that microbiome is important in skin conditions such as eczema, rosacea, acne, and many other skin conditions. Personal care products are widely used on a daily basis but it is not know how these personal care products shift the skin's microbiome. The diversity of the skin microbiome is important in the maintenance of skin equilibrium as a loss of diversity predisposes to development of skin disease.

The aim of this study is to evaluate multiple over the counter products that are used on the face daily to assess how they alter skin microbiome and diversity of microflora on skin after a week of daily treatment.

A second aim of the study is to assess how baseline diversity of microbiome are different based on self-graded skin types.

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 20-45 (limiting to females so that there is not heterogeneity with the influence of hormones. Also, females are a much larger user base of personal care products)
* Individuals in good general health
* Individuals free of any dermatological or systemic disorder, which would interfere with the results, at the discretion of the investigator
* Individuals who have participated in any other clinical studies using the same test sites (face) in the past 14 days

Exclusion Criteria:

* Individuals who have been on any topical antibiotic for the past one month or oral antibiotic therapy for the past 2 months or are currently on any antibiotic therapy
* Individuals who have history of acute or chronic disease that would likely interfere with or increase the risk on study participation at the discretion of the investigator
* Individuals with active (flaring) disease or chronic skin allergies (atopic dermatitis/eczema) or those who have recently undergone treatment for skin cancer (within the last 12 months) in the area of testing on the nose and the cheeks
* Female volunteers who are pregnant or are actively nursing
* Female volunteers who have started a new hormonal birth control agent or switched to a hormonal birth control agent within the past 60 days
* Individuals who have had any medical or cosmetic procedure, such as laser resurfacing, or plastic surgery to the test site (face) within the last 6 months. This includes botulinum toxin, dermal fillers, collagen or other similar cosmetic procedure
* Individuals who are currently using or during the past 30 days have used a retinoid such as Retin A, or other Rx/over the counter (OTC) Retinyl A or currently using or during the past 14 days have used hydroquinone (skin lightening)
* Individuals with a known history of hypersensitivity to any ingredients to the cosmetic agent that is being assessed
* Individuals with self-reported oily skin that may predispose them to acne form breakouts (at the discretion of the investigator)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females, aged 20-45
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Change in skin microflora | Baseline, 7 days
  Cotton swabs will be used to collect sample skin microbiome bacteria from the cheeks and forehead at baseline and 1 week after daily use of the intervention product. These samples will be analysed and the relative components of the microbiome will be a primary outcome.The collected measurement data will be based on a number of operational taxonomic unit (OTU).
Change in skin microbiome diversity | Baseline, 7 days
  Cotton swabs will be used to collect sample skin microbiome bacteria from the cheeks and forehead at baseline and 1 week after daily use of the intervention product. These samples will be analysed and change in diversity of the microbiome will constitute a primary outcome. The collected measurement data will be based on a number of operational taxonomic unit (OTU).

SECONDARY OUTCOMES:
Self-graded skin type | Baseline
  Types are based on the Fitzpatrick Skin Type Questionnaire, which assesses various items on Genetic Disposition, Reaction to Sun Exposure, and Tanning Habits on a score from 0-4. Skin type I corresponds to a total score of 0-7. Skin type II corresponds to a total score of 8-16. Skin type III corresponds to a total score of 17-25. Skin type IV corresponds to a total score of 25-30. Skin type V-VI correspond to a total score of over 30.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Department of Dermatology, Clinical Trials Unit, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No